CLINICAL TRIAL: NCT04788303
Title: Meals, Education, and Gardens for In-School Adolescents (MEGA) Project
Acronym: MEGA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Africa Academy for Public Health (Other); University of Dodoma (Other)
Responsible Party: Principal Investigator, Wafaie Fawzi, Professor of Nutrition, Epidemiology, and Global Health, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CNSG Project
Record Dates: First submitted 2021-02-20; First posted 2021-03-09 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Anemia
Keywords: Anemia; School garden; School lunch; Nutrition; Adolescent health
MeSH Terms: conditions — Anemia | interventions — Gardens; Educational Status

STUDY DESIGN:
Intervention Model Description: Six schools will be randomly assigned to receive the full intervention (school meal, garden, and education), partial intervention (garden and education), or control (standard of care). Community workshops will also be provided to parents of adolescents in full and partial intervention schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Full intervention (Active Comparator): Full intervention: school meal, garden, education, and community workshops
  Interventions: Other: School meal, garden, education, and community workshops
- Partial intervention (Active Comparator): Partial intervention: garden, education, and community workshops
  Interventions: Other: Garden, education, and community workshops
- Control (No Intervention): Control: standard of care

INTERVENTIONS:
Other: School meal, garden, education, and community workshops — School meal: midday meal provided at intervention schools
  School garden: garden used to grow crops (which will be used to supplement the school meal in the full intervention schools)
  Education: agriculture, nutrition, and water, sanitation, and hygiene (WASH) curriculum
  Community workshops: Led by agricultural extension workers and open to community members, the community workshops will cover nutrition messages, agricultural messages, and hands-on activities on nutrition, agriculture, and WASH.
  Other Names: Full intervention package
  Arms: Full intervention
Other: Garden, education, and community workshops — School garden: garden used to grow crops
  Education: agriculture, nutrition, and water, sanitation, and hygiene (WASH) curriculum
  Community workshops: Led by agricultural extension workers and open to community members, the community workshops will cover nutrition messages, agricultural messages, and hands-on activities on nutrition, agriculture, and WASH.
  Other Names: Partial intervention package
  Arms: Partial intervention

SUMMARY:
This purpose of this study is to assess effects of a comprehensive, school-based nutrition intervention package on anemia status, anthropometric indicators, school performance/attendance, and development indicators among adolescents, and the knowledge, attitudes, and practices of nutrition, agriculture, and WASH among parents, in Tanzania.

DETAILED DESCRIPTION:
The Meals, Education, and Gardens for In-School Adolescents (MEGA) Project aims to implement and evaluate a comprehensive, school-based nutrition intervention package among secondary schools in Dodoma, Tanzania. The intervention will include four primary components: (1) school garden, (2) school meal program, (3) agriculture, nutrition, and water, sanitation, and hygiene (WASH) education, and (4) community workshops.

This will be a cluster randomized trial with 3 arms, containing two schools each. At the beginning of the academic year, six schools will be randomized to intervention or control. Two schools will receive the full intervention package (school lunch, school garden, and education), two schools will receive the partial intervention package (school garden and education), and two schools will serve as control to receive the standard of care. Community workshops will also be provided to parents of adolescents in full and partial intervention schools.

In the full intervention schools, all adolescents will receive a midday meal, while a subset of Forms 1 or 2 adolescents will additionally participate in a school gardening program that includes nutrition, agriculture, and water, sanitation, and hygiene (WASH) education, led by selected teachers. Parents of adolescents in full intervention schools will be invited to participate in community workshops on nutrition, hygiene, and agricultural best practices, led by community Agriculture Extension Workers (AEWs).

In the partial intervention schools, Forms 1 or 2 adolescents will participate in the gardening and education components described above, but will not receive the midday meal. Parents of participating adolescents will also be invited to participate in the community workshops.

Adolescents in control schools will not receive any of these interventions but will be provided with standard of care practices at secondary schools in Dodoma. In addition, teachers in control schools will receive a hard copy of educational materials on nutrition, agriculture, and WASH to enhance their lesson plans. The intervention will take place over the course of one year.

The goal of the MEGA project is to study the effects of the integrated intervention on the nutrition and health of adolescents and their families in Tanzania. Ultimately, we aim to use the findings from this study to inform the scale-up of future school and community-based interventions to improve nutrition through training, improved crop production, and increased consumption of vegetables.

ELIGIBILITY:
INCLUSION CRITERIA:

Adolescents:

* Adolescents aged 14-17 years
* Enrolled in secondary school forms 1 or 2 at study initiation
* Member of one of the selected classes in a participating school
* Consent provided by the parent
* Assent provided by the adolescent
* Fluent in Swahili or English

Parents:

* Parent or guardian of participating adolescent
* Provides informed consent
* Fluent in Swahili or English

Teachers:

* Teacher facilitating the meal, garden, and/or education interventions
* Provides informed consent
* Fluent in Swahili or English

EXCLUSION CRITERIA:

Adolescents:

* No informed consent from parent/guardian or assent from adolescent

Parents:

* No informed consent

Teachers:

* No informed consent

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1232 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Anemia status | Up to one year
  Anemia status will be defined using the diagnostic criteria by the World Health Organization. Specifically, the following criteria will be used:
  < 12 g/dL for adolescent girls and adolescent boys aged 14 yrs and < 13 g/dL for adolescent boys aged 15-19 yrs

SECONDARY OUTCOMES:
Height | Up to one year
  Adolescent height will be measured in centimeters.
Weight | Up to one year.
  Adolescent weight will be measured in kilograms.
BMI | Up to one year
  Adolescent BMI (raw and BMI-for-age z-score based on the WHO adolescent growth standards).
Knowledge of adolescents regarding nutrition and dietary intake | Up to one year
  Adolescents' knowledge of nutrition will be assessed by questions that evaluate their levels of nutrition-related knowledge.
Attitudes of adolescents regarding nutrition and dietary intake | Up to one year
  Adolescents' attitudes of nutrition will be assessed by evaluating their preferences of food groups using Likert scales.
Practices of adolescents regarding nutrition and dietary intake | Up to one year
  Nutritional and dietary practices will be assessed using a food frequency questionnaire.
Practices of adolescents regarding water, sanitation, and hygiene | Up to one year
  Adolescents' practices of WASH will be assessed by questions that evaluate their WASH-related behaviors such as handwashing.
Educational outcomes of adolescents (school attendance) | Up to one year
  School attendance will be measured as number of school days missed per student.
Educational outcomes of adolescents (School retention) | Up to one year
  School retention will be measured as number of students who drop out of school.
Practices of WASH among parents | Up to one year
  To be assessed using questions that evaluate parents' practices on water, sanitation, and hygiene.
Home gardening practices among parents | Up to one year
  To be assessed using self-reported home gardening practice by parents.
Dietary practice among parents | Up to one year
  To be assessed using a food frequency questionnaire among parents.
Nutrition knowledge among parents | Up to one year
  To be assessed using questions that evaluate parents' knowledge on nutrition and dietary intake.

CONTACTS AND LOCATIONS:
Overall Officials: Wafaie W Fawzi, MBBS, MPH, MS, DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- University of Dodoma, Dodoma, Tanzania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang D, Katalambula LK, Modest AR, Young T, Ismail A, Mwanyika-Sando M, Tinkasimile A, Mosha D, Malero A, Vuai S, Fawzi WW. Meals, Education, and Gardens for In-School Adolescents (MEGA): study protocol for a cluster randomised trial of an integrated adolescent nutrition intervention in Dodoma, Tanzania. BMJ Open. 2022 Jul 7;12(7):e062085. doi: 10.1136/bmjopen-2022-062085. PMID 35798513